CLINICAL TRIAL: NCT05911633
Title: BioPearl™ Microspheres Loaded With Doxorubicin for the Treatment of Unresectable Hepatocellular Carcinoma (HCC): Prospective, Single Arm, Multi-center, Post-Market Clinical Follow-up (PMCF) Study
Brief Title: BioPearl™ Microspheres Loaded With Doxorubicin for the Treatment of Unresectable Hepatocellular Carcinoma (HCC)
Acronym: BIOPEARL-ONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T144E3
Record Dates: First submitted 2023-05-26; First posted 2023-06-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma Non-resectable; HCC; TACE; Chemoembolization

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Transarterial Chemo Embolization (TACE) with BioPearl™ microspheres loaded with Doxorubicin
  Interventions: Device: BioPearl™

INTERVENTIONS:
Device: BioPearl™ — TACE

SUMMARY:
The primary objective of the study is to confirm safety and technical success of BioPearl™ microspheres loaded with Doxorubicin in the treatment of unresectable hepatocellular carcinoma (HCC). The secondary objective of the study is to investigate the efficacy of BioPearl™ microspheres loaded with Doxorubicin in the treatment of subjects with unresectable HCC.

DETAILED DESCRIPTION:
This is a prospective, single arm, multi-centre, post-market clinical follow-up study to further assess safety and efficacy in 50 subjects with unresectable HCC treated with BioPearl™ microspheres loaded with Doxorubicin. All subjects will undergo clinical follow-up until disease progression and/or next treatment option, after which subjects will be followed for survival. Subjects will be followed up to a maximum of 18 months. An intermediate analysis will take place during enrollment period on safety and technical success to support regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject with HCC confirmed by histology or according to the latest applicable version of EASL (the European Association for the Study of the Liver) criteria
3. Subject with tumor(s) < 5 cm and within the up-to-7 criteria: the sum of the diameter of the largest tumor (in cm) and the number of tumors must be ≤ 7.0
4. Subject with BCLC (Barcelona Clinic Liver Cancer) Stage A or B classification who is not a candidate for curative treatment at the time of study inclusion
5. Subject with treatment failure/recurrence after a prior resection/ablation is permitted, with the exception of recurrence in the segment of a prior thermal ablation
6. WHO (World Health Organization) or ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1
7. Subject deemed treatable in one session for initial treatment
8. Normal liver or compensated cirrhosis with preserved liver function (Child-Pugh Class A)
9. Total bilirubin ≤ 2.0 mg/dl
10. Adequate bone marrow function: Hemoglobin ≥ 9g/dl, absolute neutrophil count ≥ 1.0 x 109/L, platelet count ≥ 75 x 109/L
11. Subject with no ascites or with minor ascites controlled by sodium dietary restrictions (subject receiving diuretic treatment or paracentesis is not eligible)
12. Adequate renal function: serum creatinine < 1.5 X ULN (Upper Limit of Normal)
13. Subject has provided written informed consent
14. Subjects of childbearing/reproductive potential should use adequate birth control measures, during the study treatment period until survival follow-up

Exclusion Criteria:

1. Subject previously treated with any systemic therapy for HCC
2. Subject previously treated with intra-arterial loco-regional therapy for HCC
3. Eligible for curative treatment at the time of study inclusion
4. Recurrence in the segment of a prior thermal ablation
5. Advanced liver disease: Child-Pugh's B-C class or active gastrointestinal bleeding, encephalopathy
6. Advanced tumoral disease: BCLC class C or D (vascular invasion - even segmental, extra-hepatic spread or cancer-related symptoms performance status >1)
7. History of another primary tumor. Exceptions include:

   A. Malignancy treated with curative intent ≥ 5 years before inclusion and with no known active disease

   B. Malignancy which occurred < 5 years before, not active and not expected to recur or be clinically relevant in the next 5 years
8. Subject with history of biliary tree disease or biliary dilatation
9. Portal vein thrombosis, porto-systemic shunt, hepatofugal blood flow or absent portal blood flow in the liver area to be treated
10. Contraindication to multiphasic CT and MRI (e.g. allergy to contrast media)
11. Any other contraindication for embolization procedure or Doxorubicin treatment
12. Subject is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints

    Note: Trials requiring extended follow-up for products that were investigational, but have become commercially available since then, are not considered investigational trials
13. In the Investigator's opinion subject has (a) co-morbid condition(s) that could limit the subject's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
14. Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety: by evaluating all procedural or study device related grade 3-4-5 adverse events (AEs) | Day 29
  By evaluating all procedural or study device related grade 3-4-5 adverse events (AEs) during a period of 4 weeks post initial treatment as per local investigator assessment
Technical success | Day 1
  Ability to reach near stasis in the treated tumor feeding arteries during chemoembolization procedure

SECONDARY OUTCOMES:
Tumor response rate | 18 months
  Assessed by mRECIST (modified Response Evaluation Criteria in Solid Tumors) criteria at 4 weeks and every 3 months as per local investigator assessment
Progression Free Survival (PFS) | 18 months
  Defined as time from the treatment to disease progression according to mRECIST criteria or death from any cause, whichever occurs first as per local investigator assessment
Time to progression | 18 months
  Defined as time from treatment to progression according to mRECIST criteria as per local investigator assessment
Duration of response | 18 months
  According to mRECIST as per local investigator assessment
Best response | 18 months
  Defined as best response recorded during the study according to mRECIST criteria as per local investigator assessment
Survival Rate | 18 months
  up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre Dewez, Study Director — Terumo Europe EMCD
Locations (10):
- Belgium (2):
  - CUB Hôpital Erasme, Brussels
  - UZ Leuven, Leuven
- France (3):
  - Beaujon Hospital, Clichy
  - CHU Grenobles (Hôpital Michallon), La Tronche
  - Paul-Brousse Hospital, Villejuif
- Germany (2):
  - SLK-Kliniken Heilbronn, Heilbronn
  - University Hospital Tübingen, Tübingen
- Italy (3):
  - Fondazione IRCCS Instituto Tumori, Milan
  - Fondazione Policlinico Universitario A. Gemelli, Rome
  - Città della Salute e della Scienza di Torino, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verset G, Iezzi R, Bargellini I, Bucalau AM, Pereira P, Groezinger G, Spreafico C, Maleux G. BioPearl doxorubicin microspheres for unresectable HCC: a prospective, single-arm, multicenter study: BIOPEARL-ONE. Future Oncol. 2025 Feb;21(5):557-564. doi: 10.1080/14796694.2024.2446137. Epub 2024 Dec 30. PMID 39972606